CLINICAL TRIAL: NCT04646044
Title: A Phase 1b, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Bempegaldesleukin (BEMPEG; NKTR-214) Plus Standard of Care Versus Placebo Plus Standard of Care in Adults With Mild COVID-19
Brief Title: A Placebo Controlled Trial of Bempegaldesleukin (BEMPEG; NKTR-214) With Standard of Care in Patients With Mild COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-214-34
Record Dates: First submitted 2020-11-14; First posted 2020-11-27 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Covid-19; Coronavirus Disease 2019
Keywords: BEMPEG; Bempegaldesleukin; CD122; CD122-Biased Agonist; CD122-Biased Cytokine; Coronavirus Disease; COVID-19; IL-2 receptor agonist; Lymphopenia; Mild COVID; NKTR-214; SARS-CoV-2; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — COVID-19; Lymphopenia | interventions — bempegaldesleukin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bempegaldesleukin IV + Standard of Care (Experimental)
  Interventions: Drug: Bempegaldesleukin; Drug: Standard of Care
- Placebo + Standard of Care (Placebo Comparator)
  Interventions: Drug: Standard of Care; Other: Placebo

INTERVENTIONS:
Drug: Bempegaldesleukin — Administered as an intravenous infusion
  Other Names: NKTR-214; BEMPEG
  Arms: Bempegaldesleukin IV + Standard of Care
Drug: Standard of Care — Standard of Care Treatment for COVID-19 Infection
Other: Placebo — Administered as an intravenous infusion
  Arms: Placebo + Standard of Care

SUMMARY:
The main purpose of this phase-1b, multicenter, randomized double-blind, placebo-controlled, trial is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of bempegaldesleukin (BEMPEG; NKTR-214) in combination with standard of care (SOC) in adult patients with mild COVID-19 (coronavirus disease 2019). The trial will also define the recommended phase 2 dose (RP2D) of bempegaldesleukin in patients with mild COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 years or older on the day of signing the informed consent form.
* Agrees to admission to an in-patient facility for monitoring from Days 1 to 8, inclusive.
* Symptoms of mild illness with COVID-19 without shortness of breath, dyspnea, or clinical signs indicative of more serious COVID-19.
* Laboratory confirmed SARS-CoV-2 infection within 4 days prior to the screening visit or during the 7-day screening period.
* Respiratory rate < 20 breaths per minute, heart rate < 90 beats per minute (bpm).
* Oxygen saturation by pulse oximetry > 93% on room air.
* Body mass index < 35 kg/m2.
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min.
* Alanine transaminase (ALT) or aspartate transaminase (AST) < 2 x upper limit of normal (ULN) and total bilirubin < 1.5 x ULN.
* Agrees to not participate in another clinical trial for the treatment of COVID-19 while on study unless the patient's condition has worsened and is considered to be moderate, severe, or critical by the Investigator.

Exclusion Criteria:

* Shortness of breath, hypoxia, or signs of serious lower airway disease.
* C-reactive protein, lactate dehydrogenase (LDH), or interleukin-6 (IL-6) > 1.5 x ULN.
* D-dimer or ferritin > 1.5 x ULN.
* Imminently requiring, or currently on, mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
* Systolic blood pressure < 90 mm Hg or diastolic blood pressure < 60 mm Hg.
* Evidence of acute respiratory distress syndrome (ARDS) or systemic inflammatory response syndrome (SIRS)/shock.
* Known cardiovascular history, including unstable or deteriorating cardiac disease.
* Autoimmune disease.
* History of pulmonary embolism (PE), deep vein thrombosis (DVT), or prior clinically significant venous or non-cerebrovascular accident/transient ischemic attack arterial thromboembolic event.
* Central nervous system disease or dysfunction.
* Requirement for > 2 anti-hypertensive medications.
* Unwilling to refrain from alcohol consumption from Day 1 of admission to the in-patient facility until discharge from the facility.
* Adrenal insufficiency.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (4):
- United States (4):
  - A G A Clinical Trials - HyperCore - PPDS, Hialeah, Florida
  - New Generation Medical Research, Hialeah, Florida
  - Clinical Site Partners - Winter Park - HyperCore -PPDS, Winter Park, Florida
  - SMS Clinical Research, LLC, Mesquite, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Bempegaldesleukin 0.00075 mg/kg: Bempegaldesleukin at dose of 0.00075 mg/kg was given by IV infusion as a single dose administered over 15 (± 5) minutes on Day 1
  All patients received standard of care (SOC) for COVID-19 determined by the Investigator or institution, which followed the approved prescribing guidelines in their country and institution.
- Bempegaldesleukin 0.0015 mg/kg: Bempegaldesleukin at dose of 0.0015 mg/kg was given by IV infusion as a single dose administered over 15 (± 5) minutes on Day 1
  All patients received standard of care (SOC) for COVID-19 determined by the Investigator or institution, which followed the approved prescribing guidelines in their country and institution.
- Bempegaldesleukin 0.003 mg/kg: Bempegaldesleukin at dose of 0.003 mg/kg was given by IV infusion as a single dose administered over 15 (± 5) minutes on Day 1
  All patients received standard of care (SOC) for COVID-19 determined by the Investigator or institution, which followed the approved prescribing guidelines in their country and institution.
- Placebo: Placebo control consisted of sterile normal saline solution administered at the same volume as the active administration.
  All patients received standard of care (SOC) for COVID-19 determined by the Investigator or institution, which followed the approved prescribing guidelines in their country and institution.
Period: Overall Study
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Started | 5 | 5 | 5 | 15
Completed | 5 | 4 | 4 | 15
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.5) | 31.8 (7.1) | 40.8 (12.9) | 35.6 (11.9) | 35.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 5 | 8
  Male | 3 | 5 | 4 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 4 | 13 | 24
  Not Hispanic or Latino | 2 | 1 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 4 | 5 | 4 | 14 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.2 (4.88) | 26.6 (2.03) | 27.5 (5.13) | 27.8 (4.62) | 27.6 (4.24)
Systolic Blood Pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 125.4 (7.44) | 119.2 (15.35) | 125.0 (6.28) | 122.3 (13.00) | 122.8 (11.47)
Diastolic Blood Pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 80.4 (3.21) | 77.4 (7.30) | 82.8 (5.45) | 78.1 (9.60) | 79.1 (7.81)
Pulse Rate [Mean (Standard Deviation); unit: beats/minute] | 72.8 (6.98) | 78.0 (6.52) | 79.8 (3.70) | 73.5 (9.30) | 75.2 (7.98)
Respiration Rate [Mean (Standard Deviation); unit: breaths/minute] | 15.8 (1.10) | 16.2 (0.45) | 16.6 (0.89) | 16.1 (0.52) | 16.2 (0.70)
Oxygen Saturation at Room Air [Mean (Standard Deviation); unit: %] | 97.4 (1.82) | 97.6 (0.55) | 97.8 (0.45) | 97.7 (1.33) | 97.7 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: AUC of Bempegaldesleukin [Pharmacokinetic Parameter].
Description: Area under the serum concentration-time curve (AUC) of bempegaldesleukin calculated from time 0 to 168 hours.
Time Frame: Day 1: Predose, 0.5, 24, 48, 72, 120, and 168 hours post dose.
Population: Participants with PK concentration profile to enable AUC calculation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg
Number analyzed (Participants) | 3 | 4 | 3
hr*ng/ml | 153.2 (62.5) | 997.4 (249.6) | 2704.7 (73.8)

2. Primary Outcome: Cmax of Bempegaldesleukin [Pharmacokinetic Parameter].
Description: Maximum observed serum concentration (Cmax) of bempegaldesleukin.
Time Frame: Day 1: Predose, 0.5, 24, 48, 72, 120, and 168 hours post dose.
Population: Participants with PK concentration profile to enable Cmax calculation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg
Number analyzed (Participants) | 4 | 5 | 4
ng/ml | 5.33 (135.7) | 12.67 (350.8) | 65.16 (104.1)

3. Primary Outcome: Tmax of Bempegaldesleukin [Pharmacokinetic Parameter].
Description: Time to maximum concentration of bempegaldesleukin. Cmax = maximum concentration. Tmax = time to maximum concentration.
Time Frame: Day 1: Predose, 0.5, 24, 48, 72, 120, and 168 hours post dose.
Population: Participants with PK concentration profile to enable Tmax calculation.
Measure: Median (Full Range); unit: hours
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg
Number analyzed (Participants) | 4 | 5 | 4
hours | 0.067 [0.033 to 0.417] | 0.383 [0.250 to 0.467] | 0.258 [0.083 to 18.417]

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Safety and Tolerability of bempegaldesleukin (starting at dose 0.00075 mg/kg) in combination with SOC was evaluated by incidence of Treatment-Emergent Adverse Events of Any Grade, Grade 3-4, and Grade 5 (Death).
Time Frame: Safety and tolerability were evaluated from baseline up to approximately 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
Participants
  Number of Participants with TEAEs of Any Grade | 2 | 3 | 1 | 4
  Number of Participants with TEAEs of Grade 3-4 | 0 | 0 | 0 | 0
  Number of Participants with TEAEs of Grade 5 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: Dose finding for this study was based on the assessment of DLT of bempegaldesleukin dose levels. Number and percentage of patients with any DLT were summarized by bempegaldesleukin dose level in bempegaldesleukin plus SOC treatment groups [0.00075 mg/kg, N=5; 0.0015 mg/kg, N=5; and 0.003 mg/kg, N=5] and placebo plus SOC (N=15).
  Adverse events related to study drug(s) that were defined as DLTs included the following:
  * Any Grade ≥ 3 drug-related AE.
  * Any Grade ≥ 3 drug-related laboratory abnormality that was clinically significant per the Investigator.
  * Respiratory compromise or other virus-related AE attributed to worsening COVID-19, such as severe hypoxia, cyanosis, or chest pain/pressure.
  The event was considered a DLT if it was confirmed to be at least possibly related to study drug, met any of the above definitions, and was confirmed to have occurred in a patient treated with bempegaldesleukin.
Time Frame: The DLT evaluation period was up to approximately 7 days following the bempegaldesleukin treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Percent Change From Baseline for Absolute Lymphocyte Count (ALC) by Dose/Arm.
Description: To assess the effect of bempegaldesleukin on the time course and extent of changes in absolute lymphocyte counts (ALC). Data are reported by dose and arm for Day 8 compared to baseline.
Time Frame: ALC was evaluated from baseline up to 7 days (Day 8) following the study drug administration.
Population: Analysis population included patients with both baseline and Day 8 ALC measures.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Number analyzed (Participants) | 5 | 2 | 5 | 13
Percent change from baseline | 5.85 (21.456) | 46 (NA) — According to the statistical analysis plan, if n<3, then Standard Deviation will not be calculated. | 65.82 (60.201) | -4.54 (19.663)

7. Secondary Outcome: Percentage of Patients Who Require Supplemental Oxygen.
Description: The percentage of patients requiring supplemental oxygen was evaluated as part of disease measurements to assess efficacy.
  No patient in the study required supplemental oxygen.
Time Frame: From baseline, following the administration of study drug approximately up to 30 days.
Measure: Number; unit: % of participants
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
% of participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline on the Daily Collection World Health Organization (WHO) Clinical Progression Scale, an 11-point Clinical Status Ordinal Scale.
Description: The WHO Clinical Progression Scale scores and descriptors are as follows: 0- Uninfected; no viral RNA detected; 1- Asymptomatic; viral RNA detected; 2- Symptomatic; independent; 3- Symptomatic; assistance needed; 4- Hospitalized, no oxygen therapy(a); 5- Hospitalized; oxygen by mask or nasal prongs ; 6- Hospitalized; oxygen by non-invasive ventilation or high-flow; 7- Intubation and mechanical ventilation, PaO2/FiO2 ≥ 150 or SpO2/FiO2 ≥ 200; 8- Mechanical ventilation, PaO2/FiO2 < 150 (SpO2/FiO2 < 200) or vasopressors; 9- Mechanical ventilation, PaO2/FiO2 < 150 and vasopressors, dialysis, or ECMO; 10- Death. The data are reported for Day 8 by arm. There were no scores rated 3 and higher per this scale at any timepoint.
  Abbreviations: ECMO = extracorporeal membrane oxygenation; FiO2 = fraction of inspired oxygen; PaO2 = partial pressure of arterial oxygen; SpO2 = oxygen saturation
  (a) If hospitalized for isolation only, record status as for ambulatory patient.
  Source: WHO 2020.
Time Frame: From baseline up to 7 days (Day 8) following the study drug administration.
Population: Analysis population included patients with both baseline and Day 8 scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 15
Participants
  Patients with no change from baseline | 5 | 2 | 0 | 7
  Patients with 1-point improvement | 0 | 2 | 3 | 6
  Patients with 2-point improvement | 0 | 0 | 1 | 1
  Patients with more than 2-point improvement | 0 | 0 | 0 | 0
  Patients with 1-point worsening | 0 | 0 | 1 | 1
  Patients with 2-point worsening | 0 | 0 | 0 | 0
  Patients with more than 2-point worsening | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be reported starting immediately after the patient has been administered the first dose of study drug until 30 days after the last dose of study drug, up to a maximum of approximately 40 days.
Arm/Group | Bempegaldesleukin 0.00075 mg/kg | Bempegaldesleukin 0.0015 mg/kg | Bempegaldesleukin 0.003 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 3/5 | 5/5 | 2/5 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempegaldesleukin 0.00075 mg/kg (N=5) | Bempegaldesleukin 0.0015 mg/kg (N=5) | Bempegaldesleukin 0.003 mg/kg (N=5) | Placebo (N=15)
Patients with at Least One Treatment-Emergent Adverse Event (TEAE) (General disorders) | 2 | 3 | 1 | 4 — Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event that occurs on or after the treatment dose, and treatment-emergent period is from the study dose date up to 30 days after the study dose.
Headache (Nervous system disorders) | 1 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT04646044/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04646044/SAP_001.pdf